CLINICAL TRIAL: NCT07183969
Title: The Effectiveness of Lower Extremity Strength Training on the Physical Performance of Patients With Chronic Schizophrenia With Sarcopenia.
Brief Title: The Effectiveness of Lower Extremity Strength Training
Acronym: LEST-CSchizo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chi-Tzu Shih, Ph.D. candidate, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CShih
Record Dates: First submitted 2024-07-16; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-07

CONDITIONS: Patients With Chronic Schizophrenia
Keywords: Lower extremity strength training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental groups (Experimental): 16-week lower limb muscle strength training program
  Interventions: Other: lower limb muscle strength training program
- control groups (No Intervention): received routine care

INTERVENTIONS:
Other: lower limb muscle strength training program — Each plyometric training session consists of warm-up stretching, lower limb plyometrics, and gentle stretching.
  Warm-up stretching, there are 6 movements, push the window, pull the rope, hands up, stretch from side to side, lift one foot and open and close both feet. Do 10 repetitions of each movement, 2 rounds, and keep breathing normally for a few repetitions.
  Lower Extremity Plyometrics: 3 rounds of 6 plyometrics with 1 minute of recovery time between each round. The six lower body plyometrics exercises are performed by gradually increasing the load in a manner that increases the number of seconds the exercise is held.
  Gentle Stretching: Continuous training of muscles makes them tense, stretching can lengthen muscle fibers, increase muscle elasticity, and improve blood circulation to eliminate post-training fatigue (H.K. Chen, 2022). Perform each gentle stretching movement left and right once, hold for 30 seconds each time, and keep breathing normally (no shutting up of breath).
  Arms: experimental groups

SUMMARY:
The increase in chronic schizophrenia patients with sarcopenia is currently an important healthcare issue in Taiwan and requires enhanced prevention and progress. Therefore, the purpose of this study was to understand the prevalence of sarcopenia in patients with chronic schizophrenia and to explore the effect of lower limb strength training on the physical functional performance of patients with chronic schizophrenia and sarcopenia. This study adopted a quasi-experimental design method, and the research process was divided into two stages. In the first stage, the SARC-CalF questionnaire was used to initially screen suspected chronic schizophrenia patients in a psychiatric hospital in central Taiwan. For sarcopenia cases, the skeletal muscle mass index (Skeletal Muscle Mass index) of suspected sarcopenia cases is further compared with the body composition analyzer (Inboby) to confirm the diagnosis of sarcopenia. Statistical analysis of the prevalence of sarcopenia in patients with chronic schizophrenia. In the second phase of the study, 4 chronic disease areas (two chronic disease areas for men and women) were randomly divided into experimental groups and control groups. The experimental group received a 16-week lower limb muscle strength training program, while the control group received routine care. The two groups conducted one pre-test and two post-tests, and the measurement content included physical function performance (Short Physical Performance Battery (SPPB), sarcopenia quality of life (SarQoL), and fall incidence). It is expected that the development of a set of non-pharmacological care measures will help patients in chronic psychiatric wards to become independent and slow down the progression of sarcopenia.

DETAILED DESCRIPTION:
Methods:

The purpose of this study was to investigate the effects of lower extremity muscle training on the functional performance of sarcopenia in patients with chronic schizophrenia . The study will to examine the effectiveness of a 16-week lower extremity muscle training program on the functional performance of of sarcopenia in patients with chronic schizophrenia Sample size calculation. Sample size was calculated using G*Power 3.1.9.2 software, with reference to a randomized controlled study (Nygård et al., 2023) on the integration of plyometric training into the long-term collaborative care of people with psychosis. ANOVA: Repeated measures, between factors, Effect size: 0.5, α = 0.05, Power = 0.8, 2 groups, 3 measurements per group, results showed that at least 24 cases were enrolled in each group. However, in order to increase the statistical validity and to take into account the possibility of dropout or low attendance, the default attrition rate was 25%, with 30 cases in each group. Considering that the ratio of males to females with psychosis is 1.4:1, the sample size of this study is estimated to be 40 cases in each of the experimental and control groups (24 males and 16 females in each group), making a total of 80 subjects.

Data analysis:

In this study, the data were collected and compiled, coded and entered into a computer file, and processed using the SPSS for windows version 22.0 statistical package for statistical analysis, with the significant level set at α=0.05. The data were analyzed and analyzed using the SPSS for windows version 22.0 statistical software.

Steps Based on the screening results, eight chronic wards with a high number of myasthenia gravis chronic psychosis cases were selected and divided into two groups according to gender (24 males and 16 females in each group), which were randomly assigned to the experimental and control groups by drawing lots with an opaque envelope by a non-study project staff member (a nurse practitioner supervisor). After explaining the purpose of the study and the study process to the subjects, and after the subjects had agreed to participate in the study, they were asked to sign the consent form by telephone with their family members (note the date and time of the telephone call for family members' consent). After explaining the purpose of the study and the study process to the subjects, and after the subjects had agreed to participate in the study, they were asked to sign the consent form by telephone with their family members (note the date and time of the telephone call for family members' consent).

A total of three outcome measures were assessed at pre-intervention, 8 weeks post-intervention, and 16 weeks post-intervention. In order to avoid measurement bias, the measurements in each group were performed by the same tester (facilitator).

Total of 16 weeks of lower extremity strength training was implemented in the experimental group. The training content was designed with reference to the literature and in discussion with senior psychiatric nursing staff, an ageing physical fitness instructor, and the director of the rehabilitation department, and was attempted to be taught in the community to elderly people with sarcopenia and in a chronic psychiatric ward in central China, to confirm that it was feasible to implement and that it was expected to be effective. The total number of interventions in this study was 48 (3 per week, each lasting approximately 1 hour for 16 weeks). In the week prior to the study intervention, the same professional physical fitness instructor and facilitator came to the lobby of the experimental group ward to teach and instruct the subjects on the lower limb plyometric exercises 3 times a week for 1 hour, for a total of 3 sessions. 16 weeks of the lower limb plyometric interventions were conducted by the same professional physical fitness instructor for the female ward and by the same facilitator for the male ward.

In the experimental wards, lower extremity muscle training was performed once every 3 days per week at a time slot selected by the facilitator, who assessed with the ward nursing staff the appropriateness of the day's vital signs and physical condition for performing the lower extremity training. Because of the benefits of lower extremity strength training in preventing sarcopenia and falls, after the completion of this study, the control group will be provided with instruction and guidance on lower extremity strength training maneuvers, 3 times per week for 1 hour each time, for a total of 3 times, and will be encouraged to continue to perform the exercises in their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* (1) Suitable for participation in this study as assessed by the attending physician.
* (2) After explaining the purpose of the study and the study process, family members and study subjects were asked to agree to participate in the study and to complete the consent form for signature.

Exclusion Criteria:

* (1) Those who are unable to walk unaided.
* (2) Severe structural disability that prevents the performance of lower extremity training.
* (3) Those with severe psychiatric symptoms that prevent them from concentrating and following instructions.
* (4)Participation in a lower extremity muscle training program or intervention within one year.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | baseline、8weeks、16weeks
  Chair Stand Test' Chair Stand Test、Balance tests、 Gait speed test
The Sarcopenia Quality of Life Questionnaire (SarQoL-TW) | baseline、8weeks、16weeks
  Chinese version of the Taiwan version
fall incidence | baseline、8weeks、16weeks
  medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Tsaotun Psychiatric Center,MOHW, Tsaotun, Nanton, Taiwan

IPD SHARING:
Plan to Share IPD: No
無